CLINICAL TRIAL: NCT02899611
Title: A Dose Ranging Pilot Study to Assess Intracerebroventricular (ICV) Delivery of Valproate in Subjects With Focal Seizures, With Temporal Lobe Onset With or Without Secondary Generalization
Brief Title: A Dose Ranging Pilot Study for Intracerebroventricular (ICV) Delivery of Valproate in Subjects With Temporal Seizures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cerebral Therapeutics LLC (Industry)
Collaborators: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA071976
Record Dates: First submitted 2016-09-03; First posted 2016-09-14 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid; Epilim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICV Valproate (Experimental): Patients receive a daily dose of ICV Valproate that increases from 3 mg to 60 mg (or MTD) over 8 weeks. A placebo week is randomly inserted in the dose escalation. During the placebo week, the patient receives normal saline.
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Valproate — ICV Valproate is a dilution of the commercially available Epilim product, which is a sterile intravenous (IV) formulation of Sodium Valproate.
  Other Names: Valproic acid; Depacon; Epilim

SUMMARY:
Patients with medically refractory epilepsy will be treated by intracerebroventricular (ICV) delivery of valproate using an implantable drug pump system. The dose of valproate will be escalated weekly during a blinded-evaluation period through Day 64 to determine the maximum tolerated dose (MTD). After Day 64, patients can continue for 52 weeks in the open-label evaluation period (non-blinded). .

DETAILED DESCRIPTION:
Epilepsy patients that are refractory to oral anti-epileptic drug (AED) treatment have significantly higher mortality, higher morbidity, higher economic costs and diminished quality of life compared to those who suffer from epilepsy that can be adequately controlled with medical management. Current options for refractory patients include neurosurgical brain resection, responsive neurostimulation, and vagal nerve stimulation. None of these options is satisfactory due to the low applicability of surgery for patients with poorly localized or multifocal seizures and the limited success of currently available alternative treatment options.

In this study, patients with medically refractory focal epilepsy will be treated with intracerebroventricular (ICV) administration of valproate using an implantable drug pump system. This is a dose ranging study, with a randomized, double-blind dose escalation component, to establish the dose range of ICV valproate delivery. Clinical assessments, adverse events (AEs), seizure diaries, concomitant medications, blood samples and cerebrospinal fluid (CSF) will be collected and reviewed at designated time points. Magnetic resonance imaging (MRI) and electroencephalography (EEG) will also be performed. Subjects will have their surgery, dose changes and pharmacokinetics performed in an inpatient setting.

The ICV Valproate dose will be escalated stepwise from 3 mg/day to 60 mg/day through Day 64 if tolerated, or stopped earlier upon establishment of a subject's maximum tolerated dose (MTD). The MTD for each subject will be determined based on the highest dose tolerated without experiencing a dose-limiting adverse event (AE). After establishing a subject's MTD, delivery of ICV Valproate will continue at the MTD through Day 64 of the blinded evaluation period. Subjects and assessing physicians will remain blinded to the treatment dose during the blinded evaluation period. Subjects can continue in the open-label evaluation period (non-blinded) for 52 weeks following the blinded evaluation period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 65 years old.
2. Subject does not have coagulopathy, ventricular anatomic distortion or abnormally low brain weight or significant volume loss etc. and is approved to have surgery.
3. Subject had onset of epilepsy after age 5, had normal brain development up to age 5, and has full scale IQ > 70 by testing or functional assessment.
4. Subject has brain volume which is not noted to be abnormally small due to atrophy by either the radiologist reading on MRI scan or the treating clinicians (the neurosurgeon) review of the MRI scan.
5. Subject has had confirmed epilepsy for a minimum of 1 year, with diagnosis of focal seizures with temporal lobe onset, with or without secondarily generalized seizures, as defined by the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (1981).
6. In the opinion of the investigator, subject has disabling seizures. Disabling refers to seizures that are severe enough to cause injuries, or significantly impair functional ability in domains including employment, psychosocial education and mobility.
7. Subject has had a CT or MRI of the brain to rule out progressive structural lesions.
8. Subject has had an EEG or video EEG or invasive monitoring within the past 3 yrs consistent with partial seizures (a normal interictal EEG is consistent with partial seizures)
9. Subject has previously failed at least 3 AEDs in single or combination use.
10. Subject is taking currently approved AED medication(s) (but is not on valproate or divalproex sodium) and has been on a stable dosing regimen for 1 month prior to Screening.
11. Subject has completed all investigations necessary to satisfy the PI that noninvasive therapies are not likely to be satisfactorily successful.
12. For the 3 months before informed consent an average of four or more clinically significant focal seizures of temporal lobe onset, with or without secondary generalization, per month. Only seizures with objectively visible manifestations should be counted. The subject should have no period longer than 30 days in the 3 months prior to enrollment with less than 2 seizures. Seizures of hippocampal origin are preferred if the seizure origin is known or determined from imaging and seizure localization.
13. Subject has seizures that are distinct, stereotypical events that can be reliably counted, in the opinion of the Investigator, by the subject or caregiver.
14. Subject has hearing, vision, and physical abilities adequate to perform assessments, with or without corrective aids, including keeping a seizure and medication diary during study follow-up.
15. Subject understands study procedures and has voluntarily provided signed, informed consent in accordance with institutional and local regulatory requirements.
16. Medically refractory for more than one year.
17. Needs be literate in English or native language of the country of the study enrollment to complete neuropsychological testing.
18. Subject can be reasonably expected to maintain a seizure diary alone or with the assistance of a competent individual.
19. Women of childbearing potential must be using a medically accepted method of contraception and have a negative qualitative β-human chorionic growth hormone (β-HCG) pregnancy test result from a urine or blood sample collected at Screening.

Non-childbearing potential is defined as any female who is post menopausal since the last 1 year or has had hysterectomy or bilateral oophorectomy or is surgically sterilized.

Medically accepted forms of birth control include:

1. Intrauterine device in place for at least 3 months
2. Adequate barrier methods (e.g., diaphragm and foam), or an oral contraceptive in combination with another method (e.g., spermicidal cream). An oral contraceptive alone is not considered adequate for this study.

If on hepatic inducing AEDs which could lower serum hormone levels (phenytoin, phenobarbital, primidone, carbamazepine, oxcarbazepine, topiramate, zonisamide, rufinamide, lacosamide) then an oral contraceptive must have minimum dosage equivalent to 50 µg daily of ethinyl estradiol.

Exclusion Criteria:

1. Subject has any significant neurologic disease other than epilepsy.
2. Subject has history, within 12 months prior to Screening, of repetitive seizures that cannot be counted.
3. Subject has pseudoseizures or seizures secondary to illicit drug or alcohol use, neoplasia, active CNS infection, demyelinating disease, degenerative neurological disease, progressive central nervous system disease or metabolic illness.
4. Subject has been diagnosed with partial motor, primarily generalized seizures or has been diagnosed with psychogenic or nonepileptic seizures in the preceding year.
5. Subject has had status epilepticus refractory to benzodiazepines and phenytoin within one year prior to Screening
6. Subject is currently taking neuroleptic medication for behavior control.
7. Subject is taking scheduled doses of benzodiazepines or has required, in the 3 months prior to Screening, benzodiazepine use more than 4 times per month for seizure control. One use is defined as taking up to 3 doses in a 24 hour period.
8. Subject is currently implanted with an activated DBS, or RNS device used for treatment of a neurologic or psychiatric condition.
9. Subject has VNS and the VNS stimulation parameters are not stable. Stable shall be defined such that the stimulation parameters have been changed in the last 4 months or the patient/designee is able to report "magnet swipe" during the same time period.
10. Subject is currently taking oral valproic acid or sodium divalproex.
11. Subject has refractory motor seizures.
12. Subject has had more than 10 seizures in one day or more than 300 seizures in one month within the last year.
13. Subject has known allergy to valproic acid, divalproex sodium, Epilim, or Depacon.
14. Subject has unstable depression being treated with more than 1 anti-depressant medication, or has current evidence of or history within the past 2 years of DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, and prior suicide attempt within five years. Also excluded are subjects with a history of postictal psychosis or psychosis or depression secondary to a discontinued AED.
15. Subject has had alcohol or substance abuse within the past 5 years.
16. Subject has uncontrolled Type I or Type II diabetes, hypercoagulability. Controlled diabetics for >12 months as evidenced by HbA1C <8% can be included in study based on Investigators assessment.
17. Subject has history or evidence of congestive heart failure, clinically significant peripheral edema, or anemia with a hematocrit <30%.
18. Subject has liver function tests aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at Screening ≥ 3 times the upper limit of normal, or clinically significant renal disease or insufficiency.
19. Subject has elevated (clinically significant thrombocytosis) or decreased (< 175/μL) platelet count. Subjects should not be taking aspirin or nonsteroidal anti-inflammatory drugs within the week before and week after implantation of catheter and pump.
20. Subject has abnormal prothrombin time or INR (> 14 seconds) or partial thromboplastin time (> 50 seconds).
21. Subject has, after 3 minutes in the supine position, systolic blood pressure < 90 or > 180 or pulse outside the range of 50-100 beats per minute.
22. Subject has had cancer within 3 years prior to Screening with the exception of squamous and basal cell carcinomas of the skin, and in situ carcinoma of the breast or cervix.
23. Subject is on chronic anticoagulants or, in the opinion of the Investigator, is not a suitable candidate for cranial surgery for any reason.
24. Subject has known HIV infection or known or suspected prion disease.
25. Subject has known allergies to drugs or excipients.
26. Subject is breastfeeding.
27. In the opinion of the investigator, the subject has a clinically significant or unstable medical condition (including alcohol and/or drug abuse) or a progressive CNS disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 2 months
  The ICV Valproate dose will be escalated stepwise through Day 64, if tolerated, or stopped earlier upon establishment of a subject's MTD. The MTD for each subject will be determined based on the highest dose tolerated without experiencing a dose-limiting AE.
Safety: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 14 months
  Safety will be evaluated by monitoring for adverse events (AEs) and serious adverse events (SAEs). This will be monitored using various metrics including: clinical assessments, seizure diaries, concomitant medications, blood and CSF sampling. MRI Scan, EEG and ECG will also be performed and monitored to evaluate safety.
Changes in the Number of Seizures | 14 months
  Seizure diaries will be collected, monitored and reviewed at designated time points.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | 20 months
  Peak Plasma Concentration (Cmax) will be measured for plasma and cerebrospinal fluid levels of valproate for each subject.
Pharmacokinetic Parameters 2 | 20 months
  Area Under Curve will be measured for plasma and cerebrospinal fluid levels of valproate for each subject.
Pharmacokinetic Parameters 3 | 20 months
  Half Life will be measured for plasma and cerebrospinal fluid levels of valproate for each subject.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cook M, Murphy M, Bulluss K, D'Souza W, Plummer C, Priest E, Williams C, Sharan A, Fisher R, Pincus S, Distad E, Anchordoquy T, Abrams D. Anti-seizure therapy with a long-term, implanted intra-cerebroventricular delivery system for drug-resistant epilepsy: A first-in-man study. EClinicalMedicine. 2020 May 3;22:100326. doi: 10.1016/j.eclinm.2020.100326. eCollection 2020 May. PMID 32395709